CLINICAL TRIAL: NCT05560529
Title: Dialectical Behavioral Therapy As A Therapeutic Tool In Patients With Binge Eating Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201665
Record Dates: First submitted 2022-09-24; First posted 2022-09-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Binge Eating Disorder
Keywords: Binge Eating Disorder; Ghrelin; Dialectical Behavioral Therapy
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBT (Group A) (Experimental): DBT to be applied over 20 weeks
  Interventions: Behavioral: DBT; Diagnostic Test: Plasma Ghrelin
- TAU (Group B) (Active Comparator): TAU to be applied over 20 weeks
  Interventions: Drug: TAU; Diagnostic Test: Plasma Ghrelin

INTERVENTIONS:
Behavioral: DBT — Applying DBT modules in group format over 20 weeks
  Arms: DBT (Group A)
Drug: TAU — Giving TAU (usual pharmacotherapy in BED) over 20 weeks
  Arms: TAU (Group B)
Diagnostic Test: Plasma Ghrelin — Measuring fasting plasma ghrelin pre and post treatment in both arms

SUMMARY:
Binge eating disorder (BED) is one of the recently acknowledged eating disorders, with many theories underlying its pathology whether biological or psychological. From the biological perspective, changes in plasma ghrelin were hypothesized to have a major role in developing and maintaining the disorder, while from the psychopathological perspectives, abnormalities in emotion regulation were found in many patients.

Since Dialectical Behavioral Therapy (DBT) is known to target emotion dysregulation, the main aim of this study is to assess the efficacy of DBT versus treatment as usual (TAU) in BED patients, and whether plasma ghrelin level will be affected after treatment in both arms.

DETAILED DESCRIPTION:
Binge eating disorder (BED) is one of the recently acknowledged eating disorders, with many theories underlying its pathology whether biological or psychological. From the biological perspective, changes in plasma ghrelin were hypothesized to have a major role in developing and maintaining the disorder, while from the psychopathological perspectives, abnormalities in emotion regulation were found in many patients.

Since Dialectical Behavioral Therapy (DBT) is known to target emotion dysregulation, the main aim of this study is to assess the efficacy of DBT versus treatment as usual (TAU) in BED patients, and whether plasma ghrelin level will be affected after treatment in both arms, with patients being randomly allocated in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Patients diagnosed as BED according to the Diagnostic and Statistical Manual of Mental Disorders- Fifth Version (DSM-5), after providing a written informed consent
3. Overweight or obese patients (body mass index ≥ 25), or patients with a history of overweight or obesity

Exclusion Criteria:

1. Patients with known psychotic disorders or substance use disorders
2. Patients diagnosed with current major depressive or anxiety disorders
3. Patients diagnosed with borderline personality disorder
4. Patients who are actively suicidal
5. Patients with medical conditions that can affect or alter the frequency of eating and metabolism (e.g., Thyroid disorders, Diabetes Mellitus, Malignancy)
6. Patients presenting with medical complications of BED
7. The presence of purging or compensatory behaviors
8. Current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Binge Eating Severity | 30 weeks (20 weeks intervention and 10 weeks follow up)
  measure the change in BED severity using binge eating scale, with range of scores from 0 to 46. A score of 17 is a cut-off for mild or no binge eating, while 27 or more represents severe binge eating
Emotion regulation | 30 weeks (20 weeks intervention and 10 weeks follow up)
  measure the change in emotion regulation using Difficulties in Emotion Regulation Scale. Higher scores reflect worse emotional regulation

SECONDARY OUTCOMES:
Plasma Ghrelin Level | 20 weeks
  Measure Plasma Ghrelin levels in ng/mL in both arms pre and post treatment, using enzyme-linked immunosorbent assay technique

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided